CLINICAL TRIAL: NCT00177554
Title: Phase II Trial of CHOP-R Followed by Zevalin and Rituxan in Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Biogen (Industry)
Responsible Party: Samuel Jacobs,MD, University of Pittsburgh cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI #03-005
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Drug Therapy; Radioimmunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Chemotherapy and Radioimmunotherapy — CHOP-R x 3 cycles followed by zevalin and extended rituximab

SUMMARY:
The purpose of this study is to determine the complete response rate when CHOP-R chemotherapy in followed by Zevalin in previous untreated patients with follicular lymphoma

DETAILED DESCRIPTION:
Patients with follicular lymphoma who require therapy and have been previously untreated are eligible for this non-randomized, phase II study evaluating up front therapy with CHOP-R x 3 cycles followed by zevalin and 4 additional weeks of rituxan.The complete response will be determined by combining IWC criteria and PET scanning.Secondary objectives include PET-CT conversion rate, frequency and severity of adverse events, duration of complete remission and time to next lymphoma therapy.

ELIGIBILITY:
Inclusion Criteria:

* Conformed diagnosis of follicular lymphoma, grades 1,2 or 3
* No prior chemotherapy
* No prior monoclonal antibody therapy
* Bulky or symptomatic disease, stage II-IV
* Performance status 0-2

Exclusion Criteria:

* Impaired bone marrow reserve
* Presence of CNS lymphoma
* Serious nonmalignant disease or active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Complete response rate | May 2007,May 2008, May2009, May 2010

SECONDARY OUTCOMES:
PET-CT conversion rate | May2007
Frequency and severity of adverse events | May 2007
Duration of complete response | May 2007,May 2008, May 2009, May 2010
Time to next lymphoma therapy | May 2207,May2008,May2009, May2010

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A Jacobs, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cancer Centers, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Jacobs SA, Swerdlow SH, Kant J, Foon KA, Jankowitz R, Land SR, DeMonaco N, Joyce J, Osborn JL, Evans TL, Schaefer PM, Luong TM. Phase II trial of short-course CHOP-R followed by 90Y-ibritumomab tiuxetan and extended rituximab in previously untreated follicular lymphoma. Clin Cancer Res. 2008 Nov 1;14(21):7088-94. doi: 10.1158/1078-0432.CCR-08-0529. PMID 18981007